CLINICAL TRIAL: NCT03785080
Title: Non-warfarin Oral AntiCoagulant Resumption After Gastrointestinal Bleeding in Atrial Fibrillation Patients (NOAC-GAP) - a Randomised Controlled Study
Brief Title: Non-warfarin Oral AntiCoagulant Resumption After Gastrointestinal Bleeding in Atrial Fibrillation Patients
Acronym: NOAC-GAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joseph JY SUNG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NOAC-GAP
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: gastrointestinal bleeding; stroke; thromboembolism; atrial fibrillation; NOAC
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Stroke; Thromboembolism; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- restart NOAC very early (Experimental): restart NOAC within 24 hours
  Interventions: Other: restart NOAC very early
- restart NOAC early (Active Comparator): restart NOAC at 72 - 84 hours
  Interventions: Other: restart NOAC early

INTERVENTIONS:
Other: restart NOAC very early — withhold NOAC less than 24 hours Post OGD
  Arms: restart NOAC very early
Other: restart NOAC early — withhold NOAC for 72 to 84 hours Post OGD
  Arms: restart NOAC early

SUMMARY:
Current clinical society guidelines and statements are non-specific and relatively open-ended regarding the optimal timing to restart non-warfarin oral anticoagulant (NOAC) after gastrointestinal bleeding (GIB) in patients with atrial fibrillation (AF) who require the prophylactic medication for stroke prevention. These patients are at increased risk for devastating future thromboembolic events including stroke if NOAC is not resumed promptly, whilst premature resumption of anticoagulants can result in recurrent GIB, haemorrhage, anaemia, myocardial ischaemia and infarction in those with ischaemic heart disease, and even death. However, the question as to how early a NOAC can be safely restarted after acute GIB has not been previously answered, and there remains an important knowledge gap.

DETAILED DESCRIPTION:
The effectiveness and relative safety of NOACs have been demonstrated in large international studies where reductions in the incidence of stroke in patients with AF have been reported. However, the benefits of an anticoagulant are offset by increased incident rates of bleeding including gastrointestinal bleeding (GIB) and, less commonly, intracranial bleeding, warranting careful anticoagulation management during periods when patients are susceptible to the risks for bleeding, stroke and thromboembolism.

The exact duration for withholding NOAC after acute GIB is unknown and in general, current clinical society guidelines and statements are non-specific and relatively open-ended regarding the optimal timing to restart non-warfarin oral anticoagulant (NOAC) after gastrointestinal bleeding (GIB) in patients with atrial fibrillation (AF) who require the prophylactic medication for stroke prevention. These patients are at increased risk for devastating future thromboembolic events including stroke if NOAC is not resumed, whilst premature resumption of anticoagulants can result in recurrent GIB, haemorrhage, anaemia, myocardial ischaemia and infarction in those with ischaemic heart disease, and even death.

The purpose of this study is to determine if restarting NOAC very early after endoscopic haemostasis of bleeding peptic ulcer lesions is equivalent to early resumption in AF patients in terms of safety and efficacy for prevention of recurrent bleeding freedom from GIB recurrence, while maintaining undiminished benefits in reducing incident rates of systemic thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* History of AF
* Taking any kind of NOAC at the time of index acute GIB
* Acute upper GIB (non-variceal bleeding lesions accounting for the GIB) with or without endoscopic treatment confirmed endoscopic haemostasis verified by GI specialist
* Patient or next-of-kin able to provide informed consent

Exclusion Criteria:

* Concomitant stroke (including TIA) at the time of index GIB
* Requiring bridging IV heparin therapy
* Portal hypertension
* Known bleeding diathesis
* Other conditions precluding use of NOAC at the time of randomisation

  * Pregnancy
  * Tumour bleeding
  * Antidote administration to reverse anticoagulation effect of NOACs

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
recurrent gastrointestinal bleeding | 30 days
  melaena and/or haematemesis with drop in Hb >2g/dL and confirmation of bleeding by endoscopy.

SECONDARY OUTCOMES:
recurrent gastrointestinal bleeding | 90 days
  melaena and/or haematemesis with drop in Hb >2g/dL and confirmation of bleeding by endoscopy.
Ischemic stroke or transient ischaemic attack | 30 days
  an acute episode of neurologic deficit of presumed vascular or cardioembolic origin; its presence will be confirmed by a member of the neurology service
Systemic thromboembolism | 30 days
  any clinical and/or radiographic acute stroke and/or an acute peripheral arterial thromboembolic event including acute limb ischaemia, coronary embolism and arterial thromboembolism
Death | 6 months
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Joseph SUNG, MD, Principal Investigator — CUHK
Locations (3):
- Blacktown Hospital, Blacktown, New South Wales, Australia
- Endoscopy Center, Prince of Wales Hospital, Hong Kong, Hong Kong
- National University Hospital, Singapore, Singapore